CLINICAL TRIAL: NCT01744353
Title: BrUOG 278:FOLFOX-A For Pancreatic Cancer :A Brown University Oncology Research Group Study
Brief Title: BrUOG 278: FOLFOX-A For Pancreatic Cancer A Brown University Oncology Research Group Study
Acronym: 278
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Lifespan (Other); Rhode Island Hospital (Other); Memorial Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, howard safran, Principal Investigator, Brown University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 278
Record Dates: First submitted 2012-11-26; First posted 2012-12-06 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: newly diagnosed; advanced pancreatic cancer; pancreatic cancer; metastatic pancreatic cancer; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose level 1 (Experimental): Abraxane 125 mg/m2, day 1 Oxaliplatin 85 mg/m2, day 1 leucovorin 400 mg/m2, day 1 5-FU Infusion 1200 mg/m2/ days 2 days IV infusion
  Interventions: Drug: Dose level 1
- Dose level 2/ MTD (Experimental): Abraxane 150 mg/m2, day 1 Oxaliplatin 85 mg/m2, day 1 leucovorin 400 mg/m2, day 1 5-FU Infusion 1200 mg/m2/ days 2 days IV infusion
  Interventions: Drug: Dose level 2/MTD
- Dose level 3 (Experimental): Abraxane 175 mg/m2, day 1 Oxaliplatin 85 mg/m2, day 1 leucovorin 400 mg/m2, day 1 5-FU Infusion 1200 mg/m2/ days 2 days IV infusion
  Interventions: Drug: Dose level 3

INTERVENTIONS:
Drug: Dose level 1 — Abraxane 125 mg/m2 day 1, Oxaliplatin 85 mg/m2 day 1, leuocovorin 400 mg/m2 day 1, F-FU infusion 1200 mg/m2 day x 2 days IV infusion
  Other Names: 5-FU infusion, leuocovorin, oxaliplatin, Abraxane
  Arms: Dose level 1
Drug: Dose level 2/MTD — Abraxane 150 mg/m2 day 1, Oxaliplatin 85 mg/m2 day 1, leuocovorin 400 mg/m2 day 1, F-FU infusion 1200 mg/m2 day x 2 days IV infusion
  Other Names: 5-FU infusion, leuocovorin, oxaliplatin, Abraxane
  Arms: Dose level 2/ MTD
Drug: Dose level 3 — Abraxane 175 mg/m2 day 1, Oxaliplatin 85 mg/m2 day 1, leuocovorin 400 mg/m2 day 1, F-FU infusion 1200 mg/m2 day x 2 days IV infusion
  Other Names: 5-FU infusion, leuocovorin, oxaliplatin, Abraxane
  Arms: Dose level 3

SUMMARY:
The purpose of this study is to test the safety, activity and best doses of FOLFOX-A which consists of the standard chemotherapy drugs fluorouracil, leucovorin, oxaliplatin and abraxane. Each of these drugs are currently used in pancreatic cancer.

The experimental part of the study is combining these drugs together in FOLFOX-A.

DETAILED DESCRIPTION:
More active treatments are desperately needed in pancreatic cancer. The regimen of FOLFIRINOX increases survival as compared to gemcitabine but at a cost of increased toxicity. Irinotecan is responsible for much of the toxicity of FOLFIROX but may not contribute significantly to the regimen's activity. Abraxane is a new agent in pancreatic cancer. This albumin-bound nanoparticle form of paclitaxel increases tumor accumulation of paclitaxel though binding of albumin to SPARC in pancreatic cancer stroma. The investigators therefore propose a pilot study of FOLFOX (fluorouracil, leucovorin and oxaliplatin) combined with abraxane to establish the safety and preliminary activity of FOLFOX-A. Patients with inoperable (metastatic and locally advanced) pancreatic cancer will be eligible since the primary outcome is to establish the safety of FOLFOX-A.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed pancreatic ductal adenocarcinoma.
* Metastatic or locally advanced disease.
* No prior treatment for pancreatic cancer
* Radiographically measurable disease.
* No major surgery within 4 weeks of the start of study treatment. Patients must have recovered from the side effects of any major surgery at the start of study treatment. Laparoscopy and central venous catheter placement are not considered major surgery.
* Patients with serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive FOLFOX-A
* Preexisting neuropathy > grade 1.
* No prior invasive malignancy within the prior two years. However, patients with an early stage malignancy that is not expected to require treatment in the next 2 years (such as early stage, resected breast cancer or asymptomatic prostate cancer) are eligible.
* ECOG performance status 0 or 1.
* Age ≥ 18 years of age.
* Not pregnant and not nursing. Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to beginning of treatment.
* Required Initial Laboratory Values:

  * Neutrophils ≥ 1,500/μl
  * Platelet count ≥ 100,000/μl
  * Creatinine ≤ 1.5 mg/dL -or- creatinine clearance ≥ 60 mL/min
  * Total bilirubin ≤ 1.5 x ULN
  * AST (SGOT) & ALT (SGPT) ≤ 3.0 x ULN

Exclusion Criteria:

-Patients with known brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Memorial Hospital, Pawtucket, Rhode Island
  - Rhode Island Hospital (including Newport and East Greenwich locations), Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Dose Level 1: Abraxane 125 mg/m2, day 1 Oxaliplatin 85 mg/m2, day 1 leucovorin 400 mg/m2, day 1 5-FU Infusion 1200 mg/m2/ days 2 days IV infusion
- Experimental: Dose Level 2/ MTD: Abraxane 150 mg/m2, day 1 Oxaliplatin 85 mg/m2, day 1 leucovorin 400 mg/m2, day 1 5-FU Infusion 1200 mg/m2/ days 2 days IV infusion
- Experimental: Dose Level 3: Abraxane 175 mg/m2, day 1 Oxaliplatin 85 mg/m2, day 1 leucovorin 400 mg/m2, day 1 5-FU Infusion 1200 mg/m2/ days 2 days IV infusion
Period: Overall Study
Arm/Group | Experimental: Dose Level 1 | Experimental: Dose Level 2/ MTD | Experimental: Dose Level 3
Started | 6 | 26 | 3
Completed | 6 | 26 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Dose Level 1: Drug: Dose level 1 Abraxane 125 mg/m2 day 1, Oxaliplatin 85 mg/m2 day 1, leuocovorin 400 mg/m2 day 1, F-FU infusion 1200 mg/m2 day x 2 days IV infusion
  Other Names:
  5-FU infusion, leuocovorin, oxaliplatin, Abraxane
- Experimental: Dose Level 2/ MTD: Drug: Dose level 2/MTD Abraxane 150 mg/m2 day 1, Oxaliplatin 85 mg/m2 day 1, leuocovorin 400 mg/m2 day 1, F-FU infusion 1200 mg/m2 day x 2 days IV infusion
  Other Names:
  5-FU infusion, leuocovorin, oxaliplatin, Abraxane
- Experimental: Dose Level 3: Drug: Dose level 3 Abraxane 175 mg/m2 day 1, Oxaliplatin 85 mg/m2 day 1, leuocovorin 400 mg/m2 day 1, F-FU infusion 1200 mg/m2 day x 2 days IV infusion
  Other Names:
  5-FU infusion, leuocovorin, oxaliplatin, Abraxane
- Total: Total of all reporting groups
Arm/Group | Experimental: Dose Level 1 | Experimental: Dose Level 2/ MTD | Experimental: Dose Level 3 | Total
Number analyzed (Participants) | 6 | 26 | 3 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 15 | 2 | 20
  >=65 years | 3 | 11 | 1 | 15
Age, Continuous [Mean (Full Range); unit: years] | 58.83 [35 to 70] | 63.38 [41 to 82] | 63.33 [58 to 67] | 61.85 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 1 | 16
  Male | 1 | 16 | 2 | 19
Region of Enrollment [Number; unit: participants]
  United States | 6 | 26 | 3 | 35

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Toxicities to Define MTD of FOLFOX-Abraxane (A) for Newly Diagnosed, Advanced Pancreatic Cancer.
Description: MTD (Abraxane 150 mg/m2 day 1, Oxaliplatin 85 mg/m2 day 1, leuocovorin 400 mg/m2 day 1, F-FU infusion 1200 mg/m2 day x 2 days IV infusion) was defined by protocol documented and predefined DLT's in 3 dose levels.
Time Frame: For up to 30 days post completing drug, an expected average of 6 months
Measure: Number; unit: participants
Groups:
- Experimental: Dose Level 3: Drug: Dose level 3 Abraxane 175 mg/m2 day 1, Oxaliplatin 85 mg/m2 day 1, leuocovorin 400 mg/m2 day 1, F-FU infusion 1200 mg/m2 day x 2 days IV infusion
  Other Names:
  5-FU infusion, leuocovorin, oxaliplatin, Abraxan
Arm/Group | Experimental: Dose Level 1 | Experimental: Dose Level 2/ MTD | Experimental: Dose Level 3
Number analyzed (Participants) | 6 | 26 | 3
participants | 1 | 1 | 2

2. Secondary Outcome: Response Rate (if Patient's Tumor(s)Are Progressing or Being Controlled) Following Treatment With FOLFOX-A for Patients With Newly Diagnosed, Advanced Pancreatic Cancer.
Description: Data below summarizes number of patients who experienced partial response. Partial response evaluated in this study using the international criteria proposed in the Revised Response Evaluation Criteria in Solid Tumors (RECIST) Guideline version 1.1 Response Criteria Partial Response (PR) At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: pre-drug until disease progression, whichever comes first, for an expected average of 6 months
Measure: Number; unit: participants
Arm/Group | Experimental: Dose Level 1 | Experimental: Dose Level 2/ MTD | Experimental: Dose Level 3
Number analyzed (Participants) | 6 | 26 | 3
participants | 3 | 17 | 1

ADVERSE EVENTS:
Description: Our preference is to keep as documented as it shows all toxicities experienced by this combo regimen by all patients.
Groups:
- FOLFOX- A: FOLFOX-A Dose levels -1, 1, 2, 3: Three patients will be accrued to level 1. If no dose limiting toxicities (defined in section 5.2) are observed after two cycles of treatment, then accrual to level 2 will proceed. This procedure will continue until level 3 provided that the MTD has not been reached. If a DLT is observed in one of the first 3 patients in a dose level, then accrual for that level will be expanded to 6 patients. Two or more instances of DLT in a cohort of 6 patients will result in the preceding dose level being defined as the MTD. If dose level 1 is not tolerable then dose level -1 will be investigated. Once the MTD is found, the Principal Investigator will determine which dose should be assessed futher and an additional 10 patients will be treated.
  FOLFOX-A: Three patients will be accrued to level 1. If no dose limiting toxicities (defined in section 5.2) are observed after two cycles of treatment, then accrual to level 2 will proceed. This procedure will continue un
Arm/Group | FOLFOX- A
Serious Adverse Events (participants affected / at risk) | 19/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX- A (N=35)
AKI (Investigations) | 2 (2)
anemia/HGB (Investigations) | 2 (2)
Bili (Investigations) | 2 (2)
confusion (Investigations) | 2 (2)
constipation (Investigations) | 1 (1)
Creatinine (Investigations) | 2 (2)
diarrhea (Investigations) | 2 (2)
Dizziness (Investigations) | 1 (1)
dyspnea (Investigations) | 1 (1)
fatigue (Investigations) | 1 (1)
fever (Investigations) | 3 (3)
Gout/pseuso-gout (Investigations) | 1 (1)
hypokalemia (Investigations) | 1 (1)
Hypotension (Investigations) | 3 (3)
hypoxia (Investigations) | 1 (1)
Infection (Investigations) | 7 (7)
mucositits (Investigations) | 1 (1)
muscle weakness general/M&A/malaise/generalized body aches (Investigations) | 2 (2)
Nausea (Investigations) | 2 (2)
Pain abdomen (Investigations) | 2 (2)
pain extremity (knee,hip,leg,pelvis,arm,neck,shoulder,wrist,rib,elbow, back, toe) (Investigations) | 3 (3)
Pleural effusion (Investigations) | 1 (1)
pre-syncope (Investigations) | 1 (1)
rotator cuff tear (Investigations) | 1 (1)
TIA (Investigations) | 1 (1)
Thromboemblic event (pulm embol)/DVT (Investigations) | 2 (2)
vasovagal (Investigations) | 1 (1)
vomiting (Investigations) | 1 (1)
wbc (Investigations) | 1 (1)
Colonic Obstruction (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX- A (N=35)
abdominal distention (Investigations) | 1 (1)
Allergic reaction to Oxali and overall allergic reaction (Investigations) | 4 (4)
alk phos (Investigations) | 7 (7)
alopecia (Investigations) | 4 (4)
ALT (Investigations) | 16 (16)
ANC (Investigations) | 11 (11)
anemia/HGB (Investigations) | 21 (21)
anorexia (Investigations) | 7 (7)
anxiety (Investigations) | 3 (3)
AST (Investigations) | 17 (17)
blurry vision (Investigations) | 1 (1)
BUN (Investigations) | 2 (2)
Calcium/CA (Investigations) | 5 (5)
Chills/rigors (Investigations) | 3 (3)
confusion (Investigations) | 2 (2)
constipation (Investigations) | 14 (14)
Cough (Investigations) | 6 (6)
Creatinine (Investigations) | 4 (4)
dehydration (Investigations) | 3 (3)
Depression (Investigations) | 3 (3)
diarrhea (Investigations) | 15 (15)
Dizziness (Investigations) | 3 (3)
dysgeusia (taste) (Investigations) | 3 (3)
dysuria (Investigations) | 1 (1)
dyspnea (Investigations) | 1 (1)
edema (Investigations) | 9 (9)
eye disorder- other (Investigations) | 1 (1)
fatigue (Investigations) | 23 (23)
fever (Investigations) | 5 (5)
cramping extermeties (Investigations) | 2 (2)
flatulanence (Investigations) | 1 (1)
Flushing (Investigations) | 2 (2)
Folliculitis- scalp (Investigations) | 1 (1)
GERD (Investigations) | 1 (1)
Gout/pseuso-gout (Investigations) | 1 (1)
Headache (Investigations) | 3 (3)
hearing impairment (Investigations) | 1 (1)
heartburn (Investigations) | 2 (2)
hemorrhoids (Investigations) | 1 (1)
Hiccups (Investigations) | 1 (1)
hypoalbum (Investigations) | 4 (4)
hypokalemia (Investigations) | 15 (15)
Hypotension (Investigations) | 2 (2)
Infection (Investigations) | 7 (7)
insomnia (Investigations) | 2 (2)
itchiness (head/neck) (Investigations) | 1 (1)
LDH (Investigations) | 1 (1)
Lymph (Investigations) | 8 (8)
mg (Investigations) | 1 (1)
memory impairment (Investigations) | 1 (1)
mucositits (Investigations) | 6 (6)
muscle weakness general/M&A/malaise/generalized body aches (Investigations) | 6 (6)
myositis (Investigations) | 1 (1)
Nausea (Investigations) | 24 (24)
neuropathy (Investigations) | 25 (25)
Phos (Investigations) | 1 (1)
arthritis (Investigations) | 1 (1)
Pain abdomen (Investigations) | 6 (6)
Pain bone (Investigations) | 4 (4)
Pain chest (Investigations) | 3 (3)
pain epigastric (Investigations) | 1 (1)
pain extremity (knee,hip,leg,pelvis,arm,neck,shoulder,wrist,rib,elbow, back, toe) (Investigations) | 9 (9)
post nasal drip/nasal congestion (Investigations) | 2 (2)
Renal Calculi(kidney stones) (Investigations) | 1 (1)
skin laceration (L finger) (Investigations) | 1 (1)
Skin- dry (Investigations) | 2 (2)
sodium/NA (Investigations) | 15 (15)
spasticity throat (Investigations) | 1 (1)
thrombocytopenia (Investigations) | 18 (18)
Thromboemblic event (pulm embol)/DVT (Investigations) | 4 (4)
voice alteration(hoarsness) (Investigations) | 1 (1)
vomiting (Investigations) | 5 (5)
wbc (Investigations) | 13 (13)
weight loss (Investigations) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No